CLINICAL TRIAL: NCT05608538
Title: Evaluation of Nutritional Scores as Predictive Factors of Postoperative Outcome After Pancreatic Surgery
Status: Completed | Type: Observational
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Salvatore Paiella, MD, MD, PhD, Prof., Universita di Verona
Other Study IDs: NutriPanc
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Pancreatic and Peripancreatic Tumors
Keywords: Pancreatic cancer; Pancreaticoduodenotomy; Nutritional assessment score; Malnutrition; Pancreatic surgery; Distal resection; Total resection; Oncology; Clinica trial
MeSH Terms: conditions — Pancreatic Neoplasms; Malnutrition; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients scheduled for major pancreatic surgery will be screened for malnutrition by five screening scores chosen depending on their clinical applicability. After surgery, it will be evaluated which score predicts the best complications.

DETAILED DESCRIPTION:
Patients scheduled for major pancreatic surgery (pancreaticoduodenectomy, distal resection, total resection) will be screened for malnutrition by the following screening scores: Nutritional Risk Screening Score 2002; Subjective Global Assessment; Malnutrition Universal Screening Tool; Mini Nutritional Assessment and Short Nutritional Assessment Questionnaire.

The postoperative outcome will be recorded, and the predictive value of each score will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 90 years undergoing major pancreatic resections (pancreaticoduodenectomy, distal pancreatic resection, total pancreatic resection) are eligible for inclusion. All patients are informed orally about all aspects of the trial. All conditions leading to primary pancreatic resection are eligible.

Exclusion Criteria:

* patients undergoing minor pancreatic resections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of the study consists of consecutive patients, aged between 18 and 90, that will undergo major pancreatic surgery at the General and Pancreatic Surgery Unit, Pancreas Institute, University of Verona Hospital.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of nutritional assessment score as predictive of pancreatic surgery outcomes | The nutritional assessment scores are administred between 15 and 1 day before the operation. The evaluation of outcomes ends when patient are dismissed.
  Five nutritional questionnaires are administered to each patient to assess their nutritional status and then evaluate if there is a correlation between them and the postoperative outcomes.

SECONDARY OUTCOMES:
The correlation between nutritional scores and postoperative outcomes is based on age, type of disease, possible preoperative oncological treatments, and operation technique. | The nutritional assessment scores are administred between 15 and 1 day before the operation. The evaluation of outcomes ends when patient are dismissed.
  Association of each score with postoperative outcomes depending on certain patient's characteristics:age,type of disease,operation technique (open surgery versus laparoscopy)

CONTACTS AND LOCATIONS:
Locations (1):
- General and Pancreatic Surgery Unit, Pancreas Institute, University of Verona Hospital, Verona, Italy

REFERENCES:
- [Derived] Paiella S, Secchettin E, Azzolina D, De Pastena M, Gentilini N, Trestini I, Casciani F, Sandini M, Lionetto G, Milella M, Malleo G, Gianotti L, Gregori D, Salvia R. Evaluation of five nutritional scores as predictors of postoperative outcome following pancreatic resection: A prospective, single-center study. Clin Nutr ESPEN. 2024 Oct;63:635-641. doi: 10.1016/j.clnesp.2024.07.014. Epub 2024 Jul 24. PMID 39053696